CLINICAL TRIAL: NCT04291352
Title: Thalassemic Iron Overload Cardiomyopathy is Ameliorated by Taurine Supplementation (TICATS Study)
Brief Title: Thalassemic Iron Overload Cardiomyopathy is Ameliorated by Taurine Supplementation
Acronym: TICATS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Kevin H.M. Kuo, MD, MSc, FRCPC, Principal Investigator, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 18-5613
Record Dates: First submitted 2020-02-28; First posted 2020-03-02 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Thalassemia Major
MeSH Terms: conditions — beta-Thalassemia | interventions — Taurine

STUDY DESIGN:
Intervention Model Description: Prospective, double-blind, randomized control trial. Subjects are randomized to receive either taurine or placebo in addition to their standard chelation regimen for a 12 month period.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Both taurine and placebo powder inside the capsules are a white crystalline, odorless powder. The powder is loaded into clear, vegetarian, odorless capsules. Placebo and Investigational Product capsules will be packaged in 500 cc HDPE bottles.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Taurine (Experimental): 675mg taurine four times daily
  Interventions: Dietary Supplement: Taurine
- Placebo (Placebo Comparator): placebo four times daily
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Taurine — 675mg taurine four times daily
  Arms: Taurine
Other: Placebo — placebo four times daily
  Arms: Placebo

SUMMARY:
Hypothesis: Taurine, in combination with standard iron chelation therapy, is more effective than chelation therapy alone in reducing cardiac iron overload, oxidative stress and cardiac damage in β-Thalassemia.

Protocol: Sixty subjects with transfusion dependent β-Thalassemia receiving deferasirox iron chelation therapy will be recruited and randomized in a 1:1 ratio to either (1) placebo and continuation of their iron chelation or (2) a combination of iron chelation plus taurine. Transfusion and safety visits will be scheduled monthly with clinical/biochemical assessment visits every three months. The efficacy of taurine combined with standard chelation therapy will be assessed at baseline and 12 months posttreatment by both cardiac T2*MRI, and cardiac function. The recruitment period is projected to be 12 months from initiation.

ELIGIBILITY:
Participant inclusion criteria

Participants who meet all of the following criteria will qualify for entry into the study:

1. Diagnosis of transfusion-dependent Thalassemia being followed at the RBC clinic at TGH
2. Age 18 or older
3. On a stable dose of iron chelation for >30 days. Combination iron chelation regimen is allowed in the study
4. Cardiac MRI T2* ≥8ms measured within 3 months prior to randomization.
5. Preserved left ventricular ejection fraction (LVEF) >50% as measured by cardiac MRI measured within 3 months prior to randomization.

Participant exclusion criteria

Participants who meet any of the following criteria will be excluded from the study:

1. More than 16 transfusions in the past 12 months or those who are anticipated to be on a 3 week transfusion schedule during the study period
2. Serum ferritin < 500 ng/mL at screening
3. Liver iron concentration > 40 mg/g dw as measured by liver R2 MRI (FerriScan) measured within 3 months prior to randomization
4. Signs and symptoms consistent with congestive heart failure in the opinion of the investigator
5. As a result of medical review, physical examination or screening investigations, the investigator considers the subject unfit for the study.
6. No fixed address
7. Interval advent of general contraindications to MRI.
8. Taking another investigational product within 30 days of anticipated date of randomization
9. Women who are currently pregnant or plan to become pregnant during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Cardiac iron overload | 12 months
  Differences in ratio (T2* at year 1)/(T2* at baseline) between the taurine and standard chelation therapy arm

SECONDARY OUTCOMES:
Left ventricular ejection fraction | 12 months
  Differences in LVEF between the taurine and standard chelation therapy arm
Blood taurine level | 12 months
  Differences in blood taurine level between the taurine and standard chelation therapy arm
C-reactive protein | 12 months
  Differences in CRP between the taurine and standard chelation therapy arm
Interleukin-6 | 12 months
  Differences in IL-6 between the taurine and standard chelation therapy arm
Plasma MDA | 12 months
  Differences in Plasma MDA between the taurine and standard chelation therapy arm
Reduced glutathione | 12 months
  Differences in GSH between the taurine and standard chelation therapy arm

CONTACTS AND LOCATIONS:
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Undetermined at this time